CLINICAL TRIAL: NCT00314847
Title: National Multicenter Randomized Trial, Comparing Two Treatments of Myocardial Infarction Complicated With Cardiogenic Shock: Standard Treatment vs Standard Treatment Plus ECLS (Extracorporeal Life Support)
Brief Title: Comparison of Standard Treatment Versus Standard Treatment Plus Extracorporeal Life Support (ECLS) in Myocardial Infarction Complicated With Cardiogenic Shock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped prematurely due to insufficient recruitment
Sponsor: University Hospital, Caen (Other)
Responsible Party: M. Piquemal, University Hospital of Caen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECLS
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Myocardial Infarction; Shock, Cardiogenic
Keywords: Myocardial infarction; Cardiogenic shock; Extracorporeal Life Support-Impella
MeSH Terms: conditions — Myocardial Infarction; Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): IABP, inotropic drugs, antiplatelet agents according to site habits.
- Experimental (Experimental): ECLS +/- IABP, inotropic drugs, antiplatelet agents according to site habits.
  Interventions: Device: Extra-Corporeal Life Support -Impella 2.5

INTERVENTIONS:
Device: Extra-Corporeal Life Support -Impella 2.5 — Percutaneous implantation of Impella pump for a duration of 3 days as a minimum and up to 7 days (recommended)
  Other Names: IMPELLA LP 2.5
  Arms: Experimental

SUMMARY:
Cardiogenic shock is currently the main cause of death after myocardial infarction and 50% of deaths occur within the first 48 hours. To limit the extent of the myocardial necrosis is the primary objective of the treatment in this context. The symptomatic treatment of the ventricular failure alone does not allow a reduction of mortality. The immediate prognosis is not significantly improved by the current standard of care, including early revascularisation and intra-aortic balloon counterpulsation.

In order to improve the immediate prognosis, it seems necessary to limit the irreversible myocardial lesions and the systemic inflammatory response induced by an extended myocardial infarction (complement activation, cytokines production, iNOS expression, etc.). These objectives may be reached by a more extended utilization and availability of circulatory assistance methods.

The investigators propose to compare, in a randomised multicenter study, two treatments of the myocardial infarction with cardiogenic shock among 44 patients:

Standard Treatment versus ECLS-Impella +/- standard treatment.

In June 2007, an amendment replaced the device ECMO by the use of Impella intra-thoracic pump.

This amendment has been approved by the Ethic Committee on July 7, 2007. In March 2009, a new amendment has been approved by the EC. This amendment allowed to revise the number of patients to enroll (reduced to 44) and this lead us to modify also the primary endpoint : variation of BNP levels between H0 and H24 (H0 defined as the nearest value of BNP level obtained before the randomization).Showing a more important BNP levels decrease in the experimental group compared to standard treatment group, the investigators obtain an indirect argument to show a superior efficacy of the tested strategy.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction complicated with cardiogenic shock
* Patient without contraindication to IABP or ECLS-Impella

Exclusion Criteria:

* Patient with refractory cardiogenic shock
* Reperfusion > 24 hours after the pain begins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-06; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Variation of BNP levels between H0 and H24 (Ho is defined as the nearest value of BNP level before the randomization). | one month

SECONDARY OUTCOMES:
BNP levels measured at H6, H12, H48 and H72. | one month
BNP level measured at H48 after assistance weaning. | one month
haemoglobin levels | one month
lactate levels | one month
creatinine levels | one month
Mortality at day 30 or Evolution to a refractory cardiogenic shock requiring an intra-thoracic ventricular assistance or an ECMO (ECLS-Impella group) and all types of ventricular assistance (IAPB group) or a cardiac graft within 30 days. | one month
Mortality at Day 30, at 6 months, at 1 year. | one year
Infarct size at 1 month and 4 months. | 4 months
Amines maximal dose | one month
Cardiologic treatments outside the hospital | one year
Assistance last | one month
mechanical ventilation last | one month
assistance weaning failure | one month
haemorrhagic, ischemic and septic complications. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Massetti, MD, Principal Investigator — University Hospital, Caen; Rémi Sabatier, MD, Principal Investigator — University Hospital, Caen
Locations (13):
- France (13):
  - Brest University Hospital, Brest
  - Caen University Hospital, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital de la Timone, Marseille
  - Paris Sud Cardiovascular Institute, Massy
  - Mulhouse Hospital, Mulhouse
  - Pitié-Salpétrière Hospital, Paris
  - Cochin Hospital, Paris
  - Hôpital Haut-Lévèque, Pessac
  - Hôpital Charles Nicolle, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Toulouse University Hospital, Toulouse